CLINICAL TRIAL: NCT00855036
Title: Prospective Evaluation of Blunt Renal Injury in Children
Status: Terminated | Type: Observational
Why Stopped: Will be joining a consortium study with the same protocol
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00003106; 11120119 (Other: Children's Mercy Hospital)
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-08

CONDITIONS: Renal Injury
Keywords: blunt renal injury; kidney laceration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Injury: All patients who have a discernable injury to the renal parenchyma on CT scan from blunt trauma
  Interventions: Other: Attenuated bedrest

INTERVENTIONS:
Other: Attenuated bedrest — Patients are allowed to ambulate the morning after admission and then can be discharged when eating well and pain is controlled on oral pain medication regardless of hematuria
  Other Names: Renal Laceration

SUMMARY:
The objective of this study is to evaluate the outcomes of children who have sustained blunt renal injury and to evaluate our current bed rest protocol. The variables of concern are readmission, operation, subsequent hypertension and clearance of hematuria. The specific aim of the study is to prospectively collect the clinical data of these children to validate our hospital management and to define the natural history of these lesions.

DETAILED DESCRIPTION:
The current management for blunt renal injury in children is based on level 5 evidence, which is the lowest score. Essentially, empiric decisions about therapy without physiologic rationale have been permeated through generations of teaching. Patients are therefore managed by historical opinion, borrowing some principles from spleen and liver injuries. Over the past few decades all authors have agreed that non-operative management should be followed in all these patients as almost all injuries will heal with preservation of renal function. However, as opposed to spleen and liver injuries, there are no published guidelines for a non-operative management scheme. The kidney possesses important anatomic and physiologic differences when compared to the intraperitoneal solid organs that may allow for a distinct method of management. Therefore, we conducted a retrospective review to examine the natural history of these injuries and identify potential recommendations for management (IRB 07 12-186X). In patients with isolated renal injury (n = 65), mean length of bedrest was 3.8 +/- 1.9 days resulting in a mean length of stay of 3.8 +/- 3.1 days. There were no transfusions in these patients. There were 3 patients readmitted after discharge, 2 for pain control, and one for new hematuria after discharge. There were 15 patients discharged with persistent hematuria, none of whom suffered long term sequelae. Children were released from bedrest in attending-specific manner which was a wide array of management schemes. Our data suggests the risk of significant hemorrhage from blunt renal trauma is low. Further, clearance of hematuria may not be a good marker for therapy. Therefore, a period of bedrest with serial blood and urine monitoring may not be justified, and there is clearly a role for prospective application of a single management protocol to validate at least one protocol for other institutions to follow.

In the retrospective data, we found one patient developed intermittent hypertension. However, identifying this one patient requires that the hypertension is documented in our medical record, which means we may miss those patients managed by their pediatricians. More concerning is that we may be missing patients who have hypertension. These potential patients may get well into adulthood before the hypertension is detected which is why this study is imperative to define the natural history of renal healing, quantify the risk of hypertension, and potentially identify predictors of this complication.

The management protocol currently being followed and proposed for this study will include one night of bedrest and then the patient may be ambulatory the next day. From this point, patients will be managed in the hospital until they meet general discharge criteria. Discharge criteria are adequate pain control with oral pain medications and tolerating regular diet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with blunt renal injury
* Less than 18 years of age at time of injury
* Patients without known bleeding abnormalities

Exclusion Criteria:

* Children without blunt renal injury
* Children with known bleeding abnormalities
* Patients 18 years of age and older at the time of injury
* Inability to comply with the intended follow up
* Patients with open/penetrating renal trauma

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 18 who have an identifiable renal parenchymal injury on CT after blunt trauma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Hypertension | 3 years

SECONDARY OUTCOMES:
Time to clear hematuria | 2 months
length of stay | 2 weeks
degree of injury | 1 day
complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States